CLINICAL TRIAL: NCT07050303
Title: The Effect of a Mobile Application Based on the Social Cognitive Learning Theory on Medication Adherence and Hypertension Self-Efficacy in Patients With Hypertension: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gozde Aygun (Other)
Responsible Party: Sponsor-Investigator, Gozde Aygun, PhD, Muğla Sıtkı Koçman University
Organization: Muğla Sıtkı Koçman University (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 23003474
Record Dates: First submitted 2025-01-29; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Hypertension
Keywords: Hypertension; Mobile Application; Social Cognitive Learning Theory; Public Health Nursing; Hypertension Self-Efficacy Scale; Medication Adherence Self-Efficacy Scale
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participitants (Experimental): Mobile application users
  Interventions: Other: Mobile Application Developed Based on Social Cognitive Theory
- Control (No Intervention): non-users of application

INTERVENTIONS:
Other: Mobile Application Developed Based on Social Cognitive Theory — Measuring the Benefits of a 3-Month Mobile Application Use in Hypertension Patients
  Arms: Participitants

SUMMARY:
In this study, a mobile application designed based on the Social Cognitive Theory was evaluated in middle-aged individuals with hypertension:

H1(a): A mobile application based on the Social Cognitive Theory affects medication adherence self-efficacy levels in patients with hypertension.

H0(a): A mobile application based on the Social Cognitive Theory does not affect medication adherence self-efficacy levels in patients with hypertension.

H1(b): A mobile application based on the Social Cognitive Theory affects hypertension self-efficacy levels in patients with hypertension.

H0(b): A mobile application based on the Social Cognitive Theory does not affect hypertension self-efficacy levels in patients with hypertension.

H1(c): A mobile application based on the Social Cognitive Theory affects systolic and diastolic blood pressure levels in patients with hypertension.

H0(c): A mobile application based on the Social Cognitive Theory does not affect systolic and diastolic blood pressure levels in patients with hypertension.

Participants were asked to download and use the hypertension monitoring application designed by the researcher on their phones for a period of three months. A pre-test was administered through face-to-face interviews before installing the application. After using the application for three months, a post-test was conducted using the same scales through face-to-face interviews. For the control group, the same pre-test was administered through face-to-face interviews without using the application. After three months, a post-test was again conducted via face-to-face interviews.

The researchers compared the data of the participants with those of the control group.

DETAILED DESCRIPTION:
Non-communicable diseases (NCDs) account for two-thirds of all deaths globally. Hypertension, one of the NCDs, is a major risk factor for cardiovascular disability and death, affecting a high proportion of people worldwide. In Turkey, 1 in 3 people have hypertension, and it is more common in women than in men. Smartphone users have increased since 2007, and in 2019, an estimated 3.2 billion smartphone users, or about one-third of the global population, were reported. Mobile health (mHealth) technologies can be an effective way to promote hypertension self-management. Social Cognitive Learning Theory, developed by Bandura, focuses on behavioral change and the cognitive processes that influence behavior. Hypertension is a significant health problem in both developing and developed countries, and its increasing epidemic is a serious warning for more attention to this silent disease. Instead of routine and standard care interventions applied by nurses, adopting and implementing theory and model-based, scientifically supported care interventions will significantly contribute to the professionalization of the profession. When we look at the literature, it has been determined that mobile applications for hypertension patients in Turkey are limited or insufficient, and there is no mobile application based on social cognitive theory. We believe that this research will contribute to hypertension management through a mobile-based application. NCDs like hypertension are public health problems that place a heavy burden on healthcare systems and affect the entire society. This research is unique in this respect. The aim of this study is to examine the effectiveness of a mobile application on adherence to hypertension and medication treatment, and self-efficacy perception levels in hypertension patients. The study was designed as a two-group (pre-test - post-test) randomized controlled experimental design. The population of the study consists of patients aged 40-64 who applied to the Cardiology outpatient clinics of a university hospital in Aydın province within the last year (January 1 - December 31, 2024), diagnosed with hypertension, using antihypertensive drugs, and under follow-up (n=451). G-Power analysis (G Power 3.1.9.7) was used to determine the sample size. Based on the effect size of a similar study, it was determined that 82 participants should be included in the experimental and control groups, assuming a power of 0.80, an error level of 0.05, an effect size of 0.55, and a difference of 0.80. However, assuming potential losses from the sample group, 45 participants were included in the experimental group and 45 in the control group. Participants were selected through randomized control, and stratification by age and gender was performed between the two groups. Pre-test data were collected between september 25th and october 15th, 2024, and post-test data will be collected face-to-face by the researcher in the seminar hall of Aydın Adnan Menderes Application and Research Hospital between February 1, 2025, and March 30, 2025. Socio-demographic form, Short Form of Medication Adherence Self-Efficacy Scale, and Hypertension Self-Efficacy Scale will be used as data collection tools. Measurable data, such as blood pressure, height-weight, and body mass index, will be measured and recorded by the researcher. The mobile application developed by the researcher according to the Social Cognitive Theory will be applied to the experimental group. The content of the mobile application includes sub-headings such as definition and management of high blood pressure, medication use and adherence, high blood pressure and active lifestyle, high blood pressure and healthy eating, high blood pressure and stress management, high blood pressure and weight management, and the effect of smoking and alcohol consumption on high blood pressure. The follow-up period for the experimental group is set at 3 months. The control group will continue with routine care and follow-up at the hospital. Upon completion of the study, the Hypertension Self-Efficacy Scale and Medication Adherence Self-Efficacy Scale will be administered to the experimental and control groups, and measurable data will be re-recorded. When the study is completed, the mobile application will also be introduced and made available to participants in the control group if they wish. The collected data will be evaluated using SPSS 21.0 software in a computer environment. In all statistical analyses, p<0.05 will be considered statistically significant. With the developed mobile application, the additional burden and cost of the disease on the healthcare system and healthcare professionals can be reduced, and potential complications that may arise from the disease can be prevented.

Non-communicable diseases (NCDs) account for two-thirds of all deaths globally. In 2012, it was estimated that 67% of the 56 million deaths worldwide were due to non-communicable diseases (NCDs), particularly cardiovascular diseases (42.6%), cancers (21.7%), and chronic respiratory diseases (Hyder, 2017). Hypertension (HTN) is a cardiovascular syndrome characterized by a sustained elevation of arterial blood pressure, serving as one of the major risk factors for cardiovascular diseases and a leading cause of death. Hypertension is the most important risk factor for cardiovascular disability and mortality, affecting a high proportion of people worldwide (Zhang, 2021). Hypertension is considered a significant public health problem in both developed and developing countries. Hypertension prevalence rates are 36.5% in America, 36.9% in Lebanon, 34% in Australia, and 32% in Poland (Tailakh et al., 2013; Matar et al., 2015; Hering, 2018). In Turkey, 1 in 3 people have hypertension, and it is more common in women than in men (Turkish Society of Cardiology, 2022). Hypertension treatment involves various approaches, including non-pharmacological and pharmacological methods such as lifestyle modifications, physical activity, medical nutrition therapy, and medication therapy. Non-adherence to antihypertensive medication regimens is a major cause of inadequate blood pressure control. Up to 50% of failures in blood pressure control can be attributed to this non-adherence. Studies have shown that treatment of mild to moderate hypertension can reduce the risk of stroke by 30% to 43% and myocardial infarction by 15% (Yang, 2016). Sustainable Development Goals (SDGs) aim to reduce premature deaths from NCDs by one-third by 2030 (WHO, 2022). Kılıç and Türkoğlu (2021) determined in their studies that a large proportion of hypertension patients do not regularly attend their follow-ups, and nearly half do not regularly take their antihypertensive medications. Similarly, they reported that half of the patients stopped taking medication within the first year of diagnosis, and more than half stopped after approximately five years. A study mentioned that a lack of knowledge about hypertension is one of the most important reasons for ignoring high blood pressure in society. According to the results of a hypertension prevalence study conducted in Turkey in 2012, the blood pressure control rate in hypertensive patients receiving treatment was reported as 53.9%, and the reason for this was stated to be non-adherence to treatment (Kurt, 2020).

The World Health Organization recognizes the potential of digital health interventions to achieve universal health coverage and provide quality care for individuals through the use of mobile phones, web portals, or other digital tools (WHO, 2019). Smartphone users have increased since 2007, and in 2019, an estimated 3.2 billion smartphone users, or approximately one-third of the global population, were reported. With this increase, there has also been an increase in the number of health-related applications, and as of 2018, it was estimated that approximately 50% of 3.4 billion smartphone and tablet users had downloaded health-related applications (Choi et al., 2020).

As a subset of electronic health (eHealth), mobile health (mHealth) is defined as the use of mobile devices in the delivery of healthcare services, particularly through short message service (SMS) messaging, voice calls, mobile phone applications, tablets, or wearable device applications. The use of cost-effective innovative e-Health interventions such as mHealth can help improve the prevention and control of non-communicable diseases in disadvantaged populations (Saleh et al., 2018). Medication adherence is an important component of hypertension management; however, only half of all hypertensive patients are considered adherent to treatment. Forgetting to take medication is one of the most frequently reported reasons for non-adherence (Buis et al., 2017). Mobile health technologies can be an effective way to promote hypertension self-management. Mobile health applications, such as text message reminders, are thought to be a low-cost and effective way to improve medication adherence with wide accessibility (Buis et al., 2017). Tezcan (2016) reported that the expected effects of mobile health applications include creating more health-conscious individuals and healthier lifestyles, saving 30% of time spent by healthcare professionals on accessing and analyzing information, and reducing costs due to less need for hospitalizations.

Choi et al. (2020) investigated 12 studies published in Korean databases in their research titled "Mobile Application-Based Interventions for Patients with Hypertension and Ischemic Heart Disease: A Systematic Review." Of the seven studies that measured blood pressure in hypertensive patients, five found that application-based interventions reduced blood pressure, two of the three studies showed a significant decrease in body mass index in patients, and five of the seven studies reported a significant change in medication adherence. Buis et al. (2017) reported in their research titled "Text Messaging to Increase Adherence to Hypertension Medications from Primary Care and Emergency Department Settings in African Americans: Results of Two Randomized Feasibility Studies" that text message medication reminders could be effective in hypertension treatment.

Kumar et al. (2017) analyzed the top 107 applications by querying Google Play and Apple iTunes using the search terms "hypertension" and "high blood pressure" in their content analysis research on smartphone-based applications for hypertension management. They found that 72% of the applications included a monitoring function, 22% included tools to improve medication adherence, 37% contained general information about hypertension, and 8% contained information about dietary approaches to manage hypertension. They also found that some applications could directly transfer recorded information to a doctor's office in a spreadsheet or graph format.

Social learning theory is predominantly a cognitive learning theory, and its name is also referred to as Social Learning Theory and Social Cognitive Theory. In social learning theory, indirect learning based on the observation of others' behaviors is discussed. According to this learning, called Observational Learning, people can acquire general and integrated learning patterns without the need for trial and error (Bahar, 2019). According to Bandura, the first stage of learning through observation is the triggering of learning in a social context. Accordingly, model-based learning is based on a four-stage process: Attention, Retention, Motor Reproduction, and Motivation (Delibaş and Erci, 2021). Self-Regulation Capacity refers to an individual's ability to control their own behavior. Individuals control many of their behaviors, such as how much to study, how much to sleep, what to eat, what to drink, and how to behave in society. Bandura states that in the stimulus-response system, human behavior is controlled not only by external rewards and punishments but also by the individual themselves (Sümen, 2019).

Self-efficacy (SE), which expresses an individual's belief in their ability to perform or achieve a specific task, is one of the fundamental concepts at the core of Albert Bandura's Social Learning Theory. The model emphasizes that an individual's self-efficacy perception is an important determinant in initiating and maintaining health-promoting behaviors (Bandura 1982, Karadağ et al. 2011). Self-efficacy is defined as "an individual's judgment of their capacity to achieve a certain level of performance," while self-competence is defined as "an individual's beliefs about their ability to perform significantly concerning events that will affect their life" (Bandura 1982). How people feel, think, and behave differs according to their self-efficacy levels. Individuals' self-efficacy levels can increase or decrease their motivation to take action (Bandura 1982). Individuals with a strong sense of self-efficacy tend to undertake more challenging tasks and strive to achieve their goals by setting high goals for themselves. Therefore, the level of self-efficacy can be an important determining factor in hypertension management (Dikmen et al., 2016; Kaynak, 2022; Kızılcı et al., 2015). Factors facilitating learning in Social Learning Theory are classified as vicarious reinforcement, vicarious punishment, vicarious motivation, and vicarious emotionality (Bahar, 2019).

Özpulat (2015) found in her study that motivational interviewing could be used to regulate blood pressure in hypertensive individuals, positively affect individuals' perceptions of illness, enable lifestyle changes, and increase their medication adherence and self-efficacy perceptions. Karadağ et al. (2012), in their study to determine the medication adherence self-efficacy levels of hypertension patients, found that patients had high levels of medication adherence self-efficacy and that this perception was influenced by gender and medication use habits. Gönel (2019) found that those who were knowledgeable about hypertension had higher adherence to treatment.

Hypertension is a significant health problem in both developing and developed countries, and its increasing epidemic is a serious warning for more attention to this silent disease. Instead of routine and standard care interventions applied by nurses, adopting and implementing theory and model-based, scientifically supported care interventions will significantly contribute to the professionalization of the profession. When we look at the literature, it has been determined that mobile applications for hypertension patients in Turkey are limited or insufficient, and there is no mobile application developed according to social cognitive theory. We believe that this research will contribute to hypertension management through a mobile-based application. NCDs like hypertension are public health problems that place a heavy burden on healthcare systems and affect the entire society. This research is unique in this respect.

Type of Research This research was designed as a two-group, pre-test - post-test - follow-up, randomized controlled experimental design.

Place and Time of Research The research will be conducted at Aydın Adnan Menderes Application and Research Hospital between december 1st, 2024, and March 1st, 2025.

Population and Sample of the Research The population of the study consists of patients aged 40-64 who applied to the Cardiology outpatient clinics of a university hospital in Aydın province within the last year (January 1 - December 31, 2024), diagnosed with hypertension, using at least two antihypertensive drugs, and under follow-up (n=451). The age range was determined considering the prevalence of hypertension (Turkish Society of Hypertension and Renal Diseases, 2012; TURKSTAT, 2022). G-Power analysis (G Power 3.1.9.7) was used to determine the sample size. The effect size of a similar study was used as a reference in this research (Kang, Park; 2016). In line with this, calculations indicated that 82 participants should be included in the experimental and control groups, assuming a power of 0.80, an error level of 0.05, an effect size of 0.55, and a difference of 0.80. However, assuming potential losses from the sample group, it is planned to include 45 participants in the experimental group and 45 in the control group. The sample group will be selected using a simple and stratified randomization method, utilizing a table of random numbers.

Participants will be selected through randomized control; an experimental and control (blocking) group will be formed. Stratification by age and gender will be performed between the two groups (Turkish Society of Hypertension and Renal Diseases, 2012; Lu et al. 2017; Shen et al., 2017; Yang et al., 2020).

Preliminary discussions were held with the institutional authority regarding the research, clinical physicians were informed, and verbal consent for cooperation was obtained. While forming the sample group, the researcher aimed to reach participants within a 2-month period by monitoring patients in the outpatient clinics.

Data Collection Tools Socio-demographic Form: The form prepared by the researchers consists of 14 questions based on a literature review, covering the personal characteristics of the caregivers (Özpulat, 2015; Karadağ et al., 2012; Gönel, 2019).

Short Form of Medication Adherence Self-Efficacy Scale:

The Medication Adherence Self-Efficacy Scale was developed by Ogedegbe et al. (2003) and revised by Fernandez et al. (2008). Its Turkish validity and reliability study was conducted by Hacıhasanoğlu et al. (2012). The Short Form of Medication Adherence Self-Efficacy Scale aims to determine the level of medication adherence self-efficacy in patients with hypertension. The scale consists of 13 items on a four-point Likert scale ["Not at all confident" (1), "Somewhat confident" (2), "Confident" (3), "Very confident" (4)]. The lowest score that can be obtained on the scale is 13, and the highest is 52. A high score on the scale indicates good adherence to antihypertensive treatment. The Cronbach's Alpha coefficient is 0.94 (Hacıhasanoğlu et al., 2012).

Hypertension Self-Efficacy Scale:

The Hypertension Self-Efficacy Scale was developed by Han et al. (2014) to determine the self-efficacy levels of patients with hypertension. The Hypertension Self-Efficacy Scale was adapted into Turkish by Türkoğlu and Kılıç (2021). The scale consists of 20 items on a four-point Likert scale ("not at all appropriate" (1) to "very appropriate" (4)). The lowest score that can be obtained on the scale is 20, and the highest is 80. A high score on the scale indicates an increased level of self-efficacy in hypertension. The Cronbach's alpha value of the scale is 0.91 (Türkoğlu and Kılıç, 2021).

Pilot Application The developed mobile application will be tested. The testing process, conducted by the researcher, will last one week with 10 patients (outside the sample) to identify errors related to the application and evaluate its content.

Dependent/Independent Variables Dependent variables: The dependent variables of the study are the Hypertension Self-Efficacy Scale and Medication Adherence Self-Efficacy Scale scores.

Independent variable: The mobile application developed by the researcher is the independent variable.

Inclusion Criteria for the Research Diagnosis of hypertension (at least 6 months) Using at least 2 antihypertensive medications Voluntary participation in the research Aged between 40-64 years (Turkish Society of Hypertension and Renal Diseases, 2012; TURKSTAT, 2022) Literate No mental or communication-impairing problems Not pregnant or breastfeeding Ability to use a smartphone No additional comorbid diseases (cancer, DM, etc.) Having a semi-automatic upper arm blood pressure monitor at home Exclusion Criteria for the Research Experiencing problems with internet access or mobile application usage Voluntarily withdrawing from the research during the study period Ethical Committee Approval and Permissions Before starting the research, written institutional permission will be obtained from Aydın Adnan Menderes Application and Research Hospital. Ethics committee approval from Muğla Sıtkı Koçman University Health Sciences and permission to use the Short Form of Medication Adherence Self-Efficacy Scale and the Hypertension Self-Efficacy Scale have been obtained (Hacıhasanoğlu et al., 2012; Türkoğlu and Kılıç, 2021). Additionally, the study will be registered with ClinicalTrials.gov, and a registration number will be obtained. Clinical physicians will be informed about the research. After the research is verbally explained to participants, written consent will be obtained, ensuring voluntary participation. At the end of the study, the mobile application will also be introduced and made available to participants in the control group if they wish. Participants' personal information will not be shared with anyone other than the individuals conducting the research.

Statistical Methods Statistical analysis of the data will be performed using SPSS software. Pearson Chi-Square will be used for comparing categorical variables between groups, t-test or Mann Whitney U for comparing continuous variables between two groups based on their normal distribution, One Way Anova or Kruskal Wallis H for comparisons between more than two groups, and Paired sample t-test or Wilcoxon Signed Ranks for within-group comparisons. p˂0.05 will be considered statistically significant.

Content Creation of the Mobile Application The first stage for the Mobile Application Based on Social Cognitive Learning Theory was a literature review. When creating the content of the mobile application, it is planned to utilize a video recorded by the researcher (correct blood pressure measurement) and scientific graphics and images. The content of the mobile application to be used in the research is based on Social Cognitive Learning Theory, and 7 sub-headings have been created. These are: definition and management of high blood pressure, medication use and adherence, high blood pressure and active lifestyle, high blood pressure and healthy eating, high blood pressure and stress management, high blood pressure and weight management, and the effect of smoking and alcohol consumption on high blood pressure. The sub-headings will include explanations and up-to-date information indicating the content and importance of the topics. The mobile application is planned to include a blood pressure tracking chart, medication tracking chart, reminder alarms for medication and blood pressure measurement (e.g., "Don't forget to take your medication," etc.), and informative messages to be sent to participants during the day (e.g., "Your daily salt intake should not exceed 6 grams," etc.) (Turkish Hypertension Consensus Report, 2015; Hypertension Diagnosis and Treatment in Light of Current Guidelines, 2014; Carey et al., 2018; Unger et al., 2020; Hypertension Diagnosis and Treatment Guideline, 2019; ESH/ESC Arterial Hypertension Guideline, 2018; T.C. Ministry of Health Turkish Nutrition Guide, 2022; T.C. Ministry of Health Turkish Physical Activity Guide, 2014; WHO Guideline For The Pharmacological Treatment Of Hypertension In Adults, 2022).

Evaluation of the Mobile Application Content

After the mobile application content is prepared, it is planned to evaluate the mobile application by obtaining the opinions and suggestions of five faculty members in public health nursing, one expert in educational sciences, one expert in informatics, and one expert from the dietetics and physiotherapist departments. First, the content of the mobile application, initially created in Word format, will be evaluated by experts for understandability and suitability for purpose according to the following scale:

1. Appropriate
2. Somewhat appropriate (Please explain what needs to be improved)
3. Not appropriate (What are your suggestions?) Necessary adjustments will be made to the educational material based on the opinions and suggestions of these experts, and the mobile application will be finalized.

Finalizing the Mobile Application The logo for the mobile application will be decided. Support from a software company/software engineer will be obtained to transfer the prepared content and information to the mobile platform. Based on preliminary discussions for the software budget, the mobile application is estimated to cost between 25,000 and 30,000 TL. The software budget will be covered by the researcher's personal budget.

Testing the Mobile Application The developed mobile application will be tested. The testing process, conducted by the researcher, will last one week with 10 patients (outside the sample) to identify errors related to the application and evaluate its content. Systemic problems, such as readability of font size, will be identified and rectified based on feedback from patients.

Mobile Application Usage Process After the content and design of the mobile application are planned, the link to the application will be sent to experimental group participants via WhatsApp, and they will be enabled to register and log in with member access. To ensure continuous data flow and track session durations within the mobile application, the user's mobile phone must be connected to an internet source. Data recorded by users on the system and the duration of their system usage can be monitored by the researcher through the "Patient Control Panel," and patient questions can be answered within 24 hours via online consultancy services. The mobile application will be accessible to participants in the experimental group between December 1st and March 1st, 2025.

Control Group In the control group of the study, patients will not receive mobile application usage or consultancy from the researcher during the study period. Patients in the control group are expected to continue their routine outpatient clinic follow-ups. After March 30, 2025, patients in the control group will also be able to use the mobile application if they wish.

ELIGIBILITY:
Research Inclusion Criteria:

1. Diagnosed with hypertension (for at least 6 months).
2. Currently using antihypertensive medication.
3. Voluntarily agrees to participate in the research.
4. Aged between 40-64 years (Turkish Society of Hypertension and Renal Diseases, 2012; TURKSTAT, 2022).
5. Literate.
6. No mental or communication-impairing issues.
7. Not pregnant or a breastfeeding mother.
8. Able to use a smartphone with an Android operating system.
9. No additional comorbid diseases (e.g., cancer, diabetes mellitus).
10. Has a semi-automatic upper-arm blood pressure monitor at home.

Research Exclusion Criteria:

1. Experiencing issues with internet access or mobile application usage.
2. Voluntarily withdraws from the study during the research process.
3. Uses an different operating system than Android operating system.

Ages: 41 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Medication Adherence Self-Efficacy Level in Hypertension Patients | From participation until the end-point is 3 months.
  A mobile app can influence medication adherence self-efficacy levels in hypertension patients.
Hypertension Self-Efficacy Level in Hypertension Patients | From participation until the end-point is 3 months.
  A mobile app influences hypertension self-efficacy levels in hypertension patients.

SECONDARY OUTCOMES:
systolic and diastolic blood pressure | From participation until the end-point is 3 months.
  mobile application effects systolic and diastolic blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Adile TÜMER, Assosciate Professor, Study Director — Muğla Sıtkı Koçman University
Locations (1):
- Aydın Adnan Menderes University, Aydin, Efeler, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Choi JY, Choi H, Seomun G, Kim EJ. Mobile-Application-Based Interventions for Patients With Hypertension and Ischemic Heart Disease: A Systematic Review. J Nurs Res. 2020 Oct;28(5):e117. doi: 10.1097/JNR.0000000000000382. PMID 32501962
- [Background] WHO guideline Recommendations on Digital Interventions for Health System Strengthening. Geneva: World Health Organization; 2019. Available from http://www.ncbi.nlm.nih.gov/books/NBK541902/ PMID 31162915
- [Background] Zhang Q, Huang F, Zhang L, Li S, Zhang J. The effect of high blood pressure-health literacy, self-management behavior, self-efficacy and social support on the health-related quality of life of Kazakh hypertension patients in a low-income rural area of China: a structural equation model. BMC Public Health. 2021 Jun 10;21(1):1114. doi: 10.1186/s12889-021-11129-5. PMID 34112122
- [Background] Yang S, He C, Zhang X, Sun K, Wu S, Sun X, Li Y. Determinants of antihypertensive adherence among patients in Beijing: Application of the health belief model. Patient Educ Couns. 2016 Nov;99(11):1894-1900. doi: 10.1016/j.pec.2016.06.014. Epub 2016 Jun 18. PMID 27378081
- [Background] Yang Y, Liu W, Ji X, Ma C, Wang X, Li K, Li J. Extended afternoon naps are associated with hypertension in women but not in men. Heart Lung. 2020 Jan-Feb;49(1):2-9. doi: 10.1016/j.hrtlng.2019.09.002. Epub 2019 Sep 11. PMID 31521340
- [Background] Arici M, Birdane A, Guler K, Yildiz BO, Altun B, Erturk S, Aydogdu S, Ozbakkaloglu M, Ersoz HO, Suleymanlar G, Tukek T, Tokgozoglu L, Erdem Y; Turk Kardiyoloji Derneg i (TKD); Turk Ic Hastaliklari Uzmanlik Dernegi (TIHUD); Turkiye Endokrinoloji ve Metabolizma Dernegi (TEMD); Turk Nefroloji Dernegi (TND); Turk Hipertansiyon ve Bobrek Hastaliklari Dernegi. [Turkish Hypertension Consensus Report]. Turk Kardiyol Dern Ars. 2015 Jun;43(4):402-9. doi: 10.5543/tkda.2015.16243. Turkish. PMID 26142798
- [Background] Tezcan C, (2016). Sağlığa Yenilikçi Bir Bakış Açısı: Mobil Sağlık. Yayın No: TÜSİAD-T/2016-03/575
- [Background] Sümen A. (2019). Sosyal Bilişsel Teoriye Temellendirilmiş ' Çocuğumu Güneşten Koruyorum' Programının Ebeveyn Davranışlarına Etkisi, Doktora Tezi, Akdeniz Üniversitesi Sağlık Bilimleri Enstitüsü, Antalya.
- [Background] Shen Y, Chang C, Zhang J, Jiang Y, Ni B, Wang Y. Prevalence and risk factors associated with hypertension and prehypertension in a working population at high altitude in China: a cross-sectional study. Environ Health Prev Med. 2017 Apr 4;22(1):19. doi: 10.1186/s12199-017-0634-7. PMID 29165123
- [Background] Saleh S, Farah A, Dimassi H, El Arnaout N, Constantin J, Osman M, El Morr C, Alameddine M. Using Mobile Health to Enhance Outcomes of Noncommunicable Diseases Care in Rural Settings and Refugee Camps: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2018 Jul 13;6(7):e137. doi: 10.2196/mhealth.8146. PMID 30006326
- [Background] Özpulat F. (2015). Motivasyonel Görüşmenin Hipertansif Bireylerin Özyeterlilik Algısına ve İlaç Tedavisi Uyumuna Etkisi, Hacettepe Üniversitesi Sağlık Bilimleri Enstitüsü, Doktora Tezi, Ankara.
- [Background] Matar D, Frangieh AH, Abouassi S, Bteich F, Saleh A, Salame E, Kassab R, Azar RR. Prevalence, awareness, treatment, and control of hypertension in Lebanon. J Clin Hypertens (Greenwich). 2015 May;17(5):381-8. doi: 10.1111/jch.12485. Epub 2015 Jan 24. PMID 25619545
- [Background] Lu J, Lu Y, Wang X, Li X, Linderman GC, Wu C, Cheng X, Mu L, Zhang H, Liu J, Su M, Zhao H, Spatz ES, Spertus JA, Masoudi FA, Krumholz HM, Jiang L. Prevalence, awareness, treatment, and control of hypertension in China: data from 1.7 million adults in a population-based screening study (China PEACE Million Persons Project). Lancet. 2017 Dec 9;390(10112):2549-2558. doi: 10.1016/S0140-6736(17)32478-9. Epub 2017 Nov 5. PMID 29102084
- [Background] Kurt (2020). Hipertansiyon Tanısı Alan Hastalara Verilen Öz Yönetim Desteğinin Bilgi Düzeyi, Tedaviye Uyum Ve Öz Bakım Yönetimine Etkisi. Doktora Tezi. Trakya Üniversitesi Sağlık Bilimleri Enstitüsü, Edirne.
- [Background] Kumar N, Khunger M, Gupta A, Garg N. A content analysis of smartphone-based applications for hypertension management. J Am Soc Hypertens. 2015 Feb;9(2):130-6. doi: 10.1016/j.jash.2014.12.001. Epub 2014 Dec 11. PMID 25660364
- [Background] Kaynak, G. K. Kronik hastalıklarda öz yeterlilik algısı: Türkiye'de gerçekleştirilen çalışmalar üzerine bir derleme. Oltu Beşeri ve Sosyal Bilimler Fakültesi Dergisi, 3(2), 79-86.
- [Background] Karadağ, E., Karatay, G., Akkuş, Y.(2012) Bir Aile Sağlığı Merkezine Başvuran Hipertansiyon Hastalarının İlaç Tedavisine Uyum Öz Etkililik Düzeyleri. Ege Üniversitesi Hemşirelik Fakültesi Dergisi, 28(3), 85-96.
- [Background] Hyder AA, Wosu AC, Gibson DG, Labrique AB, Ali J, Pariyo GW. Noncommunicable Disease Risk Factors and Mobile Phones: A Proposed Research Agenda. J Med Internet Res. 2017 May 5;19(5):e133. doi: 10.2196/jmir.7246. PMID 28476722
- [Background] Hacıhasanoglu, R., Gözüm, S., ve Çapık, C. (2012). Hipertansif Hastalarda İlaca Uyum Öz-etkililik Ölçegi kısa formunun Türkçe'sinin geçerliligi. Anadulu Kardiyoloji Dergisi, 12(3), 241-248.
- [Background] Gönel, P. (2019). Hastaların Hipertansiyon Bilgilerinin Tedaviye Uyum ve Öz-Etkililik Düzeylerine Etkisinin Belirlenmesi (Master's thesis, Eastern Mediterranean University (EMU)-Doğu Akdeniz Üniversitesi (DAÜ)
- [Background] Dikmen Y. Denar Y. Başan H. Filiz N.Y, Hemşirelik Öğrencilerinin Öz Etkinlik-Yeterlilik Düzeylerinin İncelenmesi. Çağdaş Tıp Dergisi 2016,6(3),206-2013
- [Background] Delibaş, L., Erci, B.(2021). Sosyal Bilişsel Kuram Temelli Eğitimle Tip 1 Diyabetli Çocukların Hastalık Yönetiminin Desteklenmesi. Turkish Journal of Family Medicine and Primary Care, 15(2), 404-413.
- [Background] Buis L, Hirzel L, Dawood RM, Dawood KL, Nichols LP, Artinian NT, Schwiebert L, Yarandi HN, Roberson DN, Plegue MA, Mango LC, Levy PD. Text Messaging to Improve Hypertension Medication Adherence in African Americans From Primary Care and Emergency Department Settings: Results From Two Randomized Feasibility Studies. JMIR Mhealth Uhealth. 2017 Feb 1;5(2):e9. doi: 10.2196/mhealth.6630. PMID 28148474
- [Background] Bandura A. Self Efficacy Mechanizm in Human Agency, American Agency. American Psychologist. 1982; 37(2): 122-147.
- [Background] Bahar B, Sosyal Öğrenme Kuramı Ve Sosyal Değişim Kuramı Perspektifinden Etik Liderlik. Balkan Sosyal Bilimler Dergisi 2019,8(16),237-242
- See also: WHO (2022) Guideline for the pharmacological treatment of hypertension in adults — https://apps.who.int/iris/bitstream/handle/10665/344424/9789240033986-eng.pdf
- See also: TÜİK HanrHalkı Bilişim Teknolojileri Kullanma Oranı — https://data.tuik.gov.tr/Bulten/Index?p=Hanehalki-Bilisim-Teknolojileri-(BT)-Kullanim-Arastirmasi-2022-45587
- See also: WHO Noncommunicable Diseases Fact Sheet — https://www.who.int/news-room/fact-sheets/detail/noncommunicable-diseases
- See also: TKD Hipertansiyon Prevelansı — https://tkd.org.tr/menu/92/hipertansiyon-gorulme-sikligi
- See also: Hipertansiyon Tanı ve Tedavi Klavuzu (2019) — https://file.temd.org.tr/Uploads/publications/guides/documents/20190527160350-2019tbl_kilavuz64f1da66bf.pdf?a=1
- See also: ''Güncel Kılavuzlar Işığında Hipertansiyon Tanı ve Tedavisi'' (2014) — https://tkd.org.tr/TKDData/Uploads/files/HTBulten.pdf